CLINICAL TRIAL: NCT04374526
Title: Early transfusIon of COVID-19 Convalescent Plasma in Elderly COVID-19 Patients to Prevent Disease Progression.
Brief Title: Early transfusIon of Convalescent Plasma in Elderly COVID-19 Patients. to Prevent Disease Progression.
Acronym: LIFESAVER
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 3205
Record Dates: First submitted 2020-05-02; First posted 2020-05-05 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2020-05

CONDITIONS: Coronavirus Disease 2019 )COVID-19)
MeSH Terms: interventions — COVID-19 Serotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Convalescent plasma (Experimental): Patients receive COVID-19 Convalescent Plasma (CCP) in addition to standard therapy
  Interventions: Biological: COVID-19 Convalescent Plasma
- Standard therapy (No Intervention): Patients receive standard therapy alone

INTERVENTIONS:
Biological: COVID-19 Convalescent Plasma — ABO matched pathogen-inactivated CCP is transfused at a dose of 200 ml/day for 3 days (days 1, 2, and 3).
  Other Names: CCP
  Arms: Convalescent plasma

SUMMARY:
Older age is an independent poor outcome predictor among COVID-19 hospitalized patients . Among 72,314 COVID-19 cases, case fatality rate (CFR) was 2.3% in total population, 8% in people aged 70 to 79, and 14.8% in those aged 80 and older. In the whole population, CFR was higher in people with comorbidities, ranging from 5-6% in persons with hypertension, chronic respiratory disease, diabetes or cancer, up to 10% in those with cardiovascular diseases. Sars-CoV-2 seems to be able to induce a functional exhaustion of specified T and NK lymphocyte subpopulations, breaking down antiviral immunity. One possible explanation is that the immune system of elderly people, might be exhausted by chronic stimulation associated with comorbidities and more susceptible to this Sars-CoV-2 effect. As a result, in these patients, the activation of the innate immune system might fail to produce an adequate adaptive response (i.e., virus-specific CD8+ T-cells). This results in persistent self-induced inflammation that eventually causes mortality.

The investigators hypothesize that transfusing convalescent plasma (containing neutralizing antibodies) at an early phase of COVID-19 infection could prevent or switch off the persistent inflammatory response elicited by the virus.

The objective of this study are:

* To demonstrate the superiority of COVID-19 convalescent plasma (CCP) plus standard therapy (ST) over ST alone
* To prevent progression of pneumonia in COVID-19 patients aged ≥65 with chronic comorbidities
* To decrease viral load
* To raise anti-SARS-CoV-2 antibody titer in recipients

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65
* pneumonia at CT scan
* PaO2/FiO2 ≥300 mmHg
* Presence of one or more comorbidities (consider the list provided in Appendix A)
* Signed informed consent

Exclusion Criteria:

* Age < 65
* PaO2/FiO2 < 300 mmHg
* pending cardiopulmonary arrest
* refusal to blood product transfusions
* Severe IgA deficiency
* any life-threatening comorbidity or any other medical condition which, in the opinion of the investigator, makes the patient unsuitable for inclusion

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2021-05-26 (Actual); Study Completion 2021-05-26 (Actual)

PRIMARY OUTCOMES:
Rate of COVID-19 progression | days 1 to 14.
  Proportion of patients without progression in severity of pulmonary disease defined as worsening of 2 points in the ordinal scale of WHO within day 14

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, RM
  - Ospedale SS Annunziata, Chieti
  - Istituto Nazionale Malattie Infettive Lazzaro Spallanzani, Rome

REFERENCES:
- [Derived] Teofili L, Landolfi R, Cingolani A, Antinori A, Vecchiet J, Sanguinetti M, Gasbarrini A, Pasciuto T, Orlando N, Lamonica S. "Early transfusion of convalescent plasma in older patients with COVID-19 to prevent disease progression: A structured summary of a study protocol for a randomised controlled trial". Trials. 2020 Oct 22;21(1):875. doi: 10.1186/s13063-020-04821-1. PMID 33092632